CLINICAL TRIAL: NCT06579482
Title: Clinical Study of Non-inferiority Between Aesculus Hippocastanum 50mg, Polygonum Acre 10mg, Smilax Pepyracea 40mg, Rutin 20mg Versus Diosmin 450mg and Hesperidin 50mg Tablets in Chronic Venous Insufficiency After 3 Months of Therapy
Brief Title: Clinical Trial of Aesculus Hippocastanum and Associations Versus Diosmina and Hesperidina in Chronic Venous Insuficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Professor, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 50635421.30000.5248
Record Dates: First submitted 2023-11-13; First posted 2024-08-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Venous Insufficiency
MeSH Terms: interventions — horse chestnut seed; Association

STUDY DESIGN:
Intervention Model Description: Randomized, non-inferiority, double-blind ,comparative study
Who Masked: Participant, Care Provider, Investigator
Masking Description: coated tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aesculus hippocastanum, Polygonum acre, Smilax Pepyracea, and Rutina (Experimental): Aesculus hippocastanum 50mg, Polygonum acre 10mg, Smilax Pepyracea 40mg, Rutina 20mg
  Interventions: Drug: Aesculus hippocastanum, and associations
- Diosmina, and Hesperidina (Active Comparator): Diosmina 450mg e Hesperidina 50mg
  Interventions: Drug: Aesculus hippocastanum, and associations

INTERVENTIONS:
Drug: Aesculus hippocastanum, and associations — combination product
  Other Names: no other intervention names

SUMMARY:
To demonstrate the clinical non-inferiority of efficacy between Aesculus hippocastanum, Polygonum acre, Smilax Pepyracea, Rutin and Diosmin 450mg and Hesperidin 50mg tablets in the improvement of lower limb symptoms assessed by means of a 100mm visual scale (VAS) over 3 months among adult patients presenting with chronic venous insufficiency of the lower limbs.

DETAILED DESCRIPTION:
Phlebotonics represent a heterogeneous group of therapeutic products of natural or synthetic origin that exhibit effects on edema and/or symptoms related to chronic venous diseaseThis class of drugs is effective in improving the symptoms of chronic venous insufficiency and in cases of hemorrhoids and for this reason they have become an established component of the therapeutic arsenal for all phases of these diseases Phlebotomics are classified into four categories: benzopyrones, saponins, other plant extracts, and synthetic drugs

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting CEAP classification from grade C0 to C3 in the evaluation of venous disease of the lower limbs
2. Clinical symptoms of chronic venous insufficiency of the lower limbs, defined by the 100mm visual scale performed by the patient between 20mm and 60mm in the most symptomatic lower limb.
3. For female patients of reproductive age, not pregnant or breastfeeding, using reliable contraceptives.
4. Patient read, understood, signed and dated the free and informed consent form

Exclusion Criteria:

1. Treatment with compression stockings within 2 months of study inclusion date
2. Treatment with venotonics within 2 months of the date of inclusion in the study
3. Women of reproductive age who are pregnant or breastfeeding, or who do not wish to use contraception during the study period.
4. Known allergy or hypersensitivity to any component of the study drug
5. Known significant laboratory abnormality
6. CEAP Grade Assessment of level 4, 5, or 6.
7. Patient with venous disease requiring intravenous chemical surgery/sclerotherapy
8. Patient presenting with a painful pathology in addition to venous pain in the lower limbs 9. Patient with a history of thrombosis or thromboembolic disease within 6 months of the date of inclusion in the study

10. Patient with a change in general condition that is incompatible with his/her participation in the study 11. Patient who wishes to become pregnant within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
visual analogic scale | 3 months
  A 100 mm VAS (visual analogic scale) is marked from 0 (absence of venous symptoms) up to 100 (maximum symptomatic venous manifestations) by the patient (higher scores means a worse outcome). It is fulfilled by the patient him- or herself, under the physician's watch. VAS is meant to globally evaluate lower limbs venous symptomatology (heavy legs, painful legs, fatigued legs, deambulation limitations, swollen sensation and/or lower limbs tension).

SECONDARY OUTCOMES:
Oral acceptability by the patient through the use of a visual analogic scale | 3 months
  A 100 mm VAS (visual analogic scale) is marked from 0 (easy swallowing) up to 100 (very difficult to swallow) by the patient (higher scores means a worse outcome). It is fulfilled under by the patient him- or herself under the physician's watch.
Quality of life as measured by a specific chronic venous insufficiency questionnaire | 3 months
  CIVIQ-10 (chronIc venous insufficiency quality of life questionnaire) is a questionnaire composed of 20 scored items (on a 4 point scale) that inform on the capacity of the patient of coping with daily routine tasks, regarding their lower limbs venous competence. The higher the score, the better the clinical outcome.
Medical tolerability to tested drugs as measured by the investigator | 3 months
  Tolerability will be a measure of the nature and quantity of adverse clinical and lab reactions related to study drugs.
Patient's satisfaction to study medications | 3 months
  This endpoint regards to the medication's efficacy as perceived by the patient and graduated as: "insufficient", "acceptable", "good", or "very good".
Physician's satisfaction to study medications | 3 months
  This endpoint regards to the medication's efficacy as perceived by the investigating physician and graduated as: "insufficient", "acceptable", "good", or "very good".

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Nunes, Professor, Principal Investigator — Fundação Educacional Serra dos Órgãos
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson AG, Scholefield JH. Management of haemorrhoids. BMJ. 2008 Feb 16;336(7640):380-3. doi: 10.1136/bmj.39465.674745.80. No abstract available. PMID 18276714
- [Background] Belczak SQ, Sincos IR, Campos W, Beserra J, Nering G, Aun R. Veno-active drugs for chronic venous disease: A randomized, double-blind, placebo-controlled parallel-design trial. Phlebology. 2014 Aug;29(7):454-60. doi: 10.1177/0268355513489550. Epub 2013 May 16. PMID 23761871
- [Background] Criqui MH, Jamosmos M, Fronek A, Denenberg JO, Langer RD, Bergan J, Golomb BA. Chronic venous disease in an ethnically diverse population: the San Diego Population Study. Am J Epidemiol. 2003 Sep 1;158(5):448-56. doi: 10.1093/aje/kwg166. PMID 12936900
- [Background] Kecmanovic D, Pavlov M, Ceranic M, Sepetkovski A, Kovacevi P, Stamenkovic A. [PHLEBODIA (diosmine): a role in the management of bleeding nonprolapsed hemorrhoids]. Acta Chir Iugosl. 2005;52(1):115-6. doi: 10.2298/aci0501115k. Serbian. PMID 16119324
- [Background] Lafuma A, Fagnani F, Peltier-Pujol F, Rauss A. [Venous disease in France: an unrecognized public health problem]. J Mal Vasc. 1994;19(3):185-9. French. PMID 7798803
- [Background] Nicolaides AN, Allegra C, Bergan J, Bradbury A, Cairols M, Carpentier P, Comerota A, Delis C, Eklof B, Fassiadis N, Georgiou N, Geroulakos G, Hoffmann U, Jantet G, Jawien A, Kakkos S, Kalodiki E, Labropoulos N, Neglen P, Pappas P, Partsch H, Perrin M, Rabe E, Ramelet AA, Vayssaira M, Ioannidou E, Taft A. Management of chronic venous disorders of the lower limbs: guidelines according to scientific evidence. Int Angiol. 2008 Feb;27(1):1-59. No abstract available. PMID 18277340
- [Background] Rabe E, Guex JJ, Puskas A, Scuderi A, Fernandez Quesada F; VCP Coordinators. Epidemiology of chronic venous disorders in geographically diverse populations: results from the Vein Consult Program. Int Angiol. 2012 Apr;31(2):105-15. PMID 22466974
- [Background] Ruckley CV. Socioeconomic impact of chronic venous insufficiency and leg ulcers. Angiology. 1997 Jan;48(1):67-9. doi: 10.1177/000331979704800111. PMID 8995346
- [Background] Perera N, Liolitsa D, Iype S, Croxford A, Yassin M, Lang P, Ukaegbu O, van Issum C. Phlebotonics for haemorrhoids. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD004322. doi: 10.1002/14651858.CD004322.pub3. PMID 22895941